CLINICAL TRIAL: NCT02378337
Title: Defining PET / CT Protocols With Optimized F18-FDG (Fluorodeoxyglucose) Dose, Focusing on Reduced Radiation Dose and Improved Image Quality
Acronym: pet-ct
Status: Completed | Type: Observational
Sponsor: Hospital Sao Rafael (Other)
Responsible Party: Principal Investigator, Milena Botelho Pereira Soares, PhD, Hospital Sao Rafael
Other Study IDs: 27558714.4.0000.0048
Record Dates: First submitted 2015-02-13; First posted 2015-03-04 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Malignant Neoplasm of Breast; Hodgkin Disease; Non-Hodgkin Lymphoma, Follicular (Nodular); Malignant Neoplasm of Bronchus and Lung; Malignant Neoplasm of Colon; Secondary Neoplasm Malignant and Unspecified Lymph Nodes; Malignant Melanoma of the Skin; Malignant Neoplasm of Small Intestine
MeSH Terms: conditions — Breast Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective development cohort: A total of 85 18F-FDG-PET adult studies were gathered over a 3-month period and retrospectively evaluated.
  Interventions: Other: Image quantify
- Prospective validation cohort: To verify the application of methodology in clinical routine, we conducted a second phase of the study prospectively in 250 subjects (phase 2) using inclusion and exclusion criteria of the retrospective study (phase 1).
  Interventions: Other: Image quantify

INTERVENTIONS:
Other: Image quantify — Will be observed all patients who perform PET / CT examinations, independent of clinical indication, in nuclear medicine at Hospital Sao Rafael. Those who show interest in participating in the study, will be provided free and informed consent form (ICF) for your appreciation. This evaluation will serve for analysis and quantification of PET-CT images.

SUMMARY:
Identify the best combination of predictive variables that influence ionizing radiation dose and improved image quality through analysis and quantification of PET-CT images in simulators and patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers;
* Both genders;
* Age over 18 years;
* Clinical indication for PET-CT scan.

Exclusion Criteria:

* Pregnant women;
* Patients who have lesions in the liver metabolically active whether primary or metastatic;
* Patients with movement difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Will be observed all patients who perform PET / CT examinations, independent of clinical indication, in nuclear medicine at Hospital Sao Rafael. Those who show interest in participating in the study, will be provided free and informed consent form (ICF) for your appreciation. This evaluation will serve for analysis and quantification of PET-CT images.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Correlation of body weight with the variation coefficient (image noise). | 360 seconds
  The image noise will be measured by VOI (Volume Of Interest) in the images. The units of measure will be kilograms (kg) for body weight, and percentage for the variation coefficient.

SECONDARY OUTCOMES:
Correlation of dose-regimen with the variation coefficient (image noise). | 360 seconds
  The dose-regimen will be calculated based on radiation dose and body surface. The image noise will be measured by VOI (Volume Of Interest) in the images. The units of measure will be MegaBecquerel per kilogram (MBq/kg) for dose-regimen, and percentage for the variation coefficient.
Correlation of acquisition protocol time with the variation coefficient (image noise). | 360 seconds
  Images will be acquired every 30 seconds until a maximum of 360 seconds. The image noise will be measured by VOI (Volume Of Interest) in the images. The units of measure will be seconds for the acquisition time, and percentage for the variation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Milena BP Soares, PhD, Principal Investigator — Hospital São Rafael; Vinicius O Menezes, BSc, Study Chair — Hospital São Rafael; Marcos AD Machado, BSc, Study Chair — Hospital São Rafael; Cleiton C Queiroz, BSc, Study Chair — Hospital São Rafael; Mauro Namias, MSc, Study Chair — Fundacion Centro Diagnostico Nuclear
Locations (1):
- Hospital Sao Rafael, Salvador, Estado de Bahia, Brazil